CLINICAL TRIAL: NCT02094833
Title: Immunogenicity and Safety of Sanofi Pasteur's DTaP-IPV-Hep B-PRP~T Combined Vaccine at 2, 4, and 6 Months of Age Versus Sanofi Pasteur's DTaP IPV//PRP~T Combined Vaccine at 2, 4, and 6 Months of Age + Hep B Vaccine at 1 and 6 Months of Age, in South Korean Infants Primed With Hep B at Birth
Brief Title: DTaP-IPV-Hep B-PRP~T Combined Vaccine Versus DTaP-IPV//PRP~T Combined Vaccine + Hep B Vaccine in Hep B Primed Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L31; U1111-1127-6896 (Other: WHO)
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Haemophilus Influenzae Type b Infection; Poliomyelitis; Hepatitis B
Keywords: Diphtheria; Tetanus; Pertussis; Haemophilus influenzae type b infection; Hepatitis B; DTaP-IPV-Hep - PRP-T vaccine
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Haemophilus Infections; Poliomyelitis; Hepatitis B | interventions — Hepatitis B Vaccines; Pentavac; Euvax-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Participants will receive 3 injections of the study vaccine (DTaP-IPV-Hep B-PRP~T combined vaccine) at 2, 4, and 6 months of age
  Interventions: Biological: DTaP-IPV-Hep B-PRP~T combined vaccine
- Group B (Active Comparator): Participants will receive 2 injections of monovalent Hep B vaccine (Euvax B®) at age 1 and 6 months and 3 injections of DTaP IPV//PRP~T vaccine (Pentaxim™) at age 2, 4, and 6 months
  Interventions: Biological: DTaP-IPV//PRP~T and Hepatitis B vaccine

INTERVENTIONS:
Biological: DTaP-IPV-Hep B-PRP~T combined vaccine — 0.5 mL, Intramuscular
  Arms: Group A
Biological: DTaP-IPV//PRP~T and Hepatitis B vaccine — 0.5 mL, Intramuscular
  Other Names: Pentaxim™; Euvax B®
  Arms: Group B

SUMMARY:
The aim of this study is to evaluate the immunogenicity and safety of a novel DTaP-IPV-Hep B-PRP~T fully liquid combined hexavalent vaccine (study vaccine) administered at 2, 4, and 6 months of age compared to Sanofi Pasteur's DTaP-IPV//PRP~T combined vaccine (Pentaxim™) given at 2, 4, and 6 months of age and Hep B vaccine (Euvax B®) given at 1 and 6 months of age in South Korean infants that received a birth dose of Hep B and born to mothers documented to be serum anti-HBs Ag negative.

Primary Objective

* To demonstrate the non-inferiority in terms of seroprotection (Diphtheria, Tetanus, poliovirus types 1, 2, and 3, PRP-T, Hep B) and vaccine response for pertussis antigens (pertussis toxoid [PT] and filamentous haemagglutinin [FHA]) of Group A versus Group B, one month after the third dose of combined vaccines.

Secondary Objectives:

* To further study the immunogenicity of the two vaccination schemes, before the first dose and one month after the last dose of vaccines.
* To study the safety after each and any dose of vaccines administered in the two vaccination schemes

DETAILED DESCRIPTION:
Study participants who received a first dose of recombinant Hep B vaccine at birth will receive either DTaP-IPV-Hep B-PRP~T combined vaccine at 2, 4, and 6 months of age + 3 doses of Hep B vaccine or Hep B vaccine (Euvax B®) at 1 and 6 months of age and DTaP IPV//PRP~T combined vaccine (Pentaxim™) at 2, 4, and 6 months of age, according to the official vaccination schedule for Hep B, DTaP, poliovirus, and Hib vaccinations in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 40 days on the day of the first study visit
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative
* Participant and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures
* Born to known hepatitis B surface antigen (HBsAg) seronegative mother (documented laboratory result of HBsAg assay from the maternal blood sample is available)
* Have received one documented dose of Hep B vaccine at birth according to the national recommendations.

Exclusion Criteria:

* Participation in the 4 weeks preceding the trial inclusion or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding any trial vaccination (except Bacille Calmette Guerin (BCG) vaccine) or planned receipt of any vaccine in the 8 days following any trial vaccination
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B (except the dose of Hep B vaccine given at birth) diseases or Haemophilus influenzae type b infection with either the trial vaccine or another vaccine
* Past or current receipt of immune globulins, blood or blood-derived products or planned administration during the trial
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, since birth; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks since birth)
* Known personal or maternal history of Human Immunodeficiency Virus (HIV) or hepatitis C seropositivity
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, or Haemophilus influenzae type b infection, confirmed either clinically, serologically, or microbiologically
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Known thrombocytopenia, as reported by the parent/legally acceptable representative
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* In an emergency setting, or hospitalized involuntarily
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study
* History of seizures.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with anti-Diphtheria antibody concentrations ≥ 0.01 International Units (IU)/mL | 1 month post third vaccination
  Anti-Diphtheria antibodies will be measured by a toxin neutralization test
Number of participants with anti-Tetanus antibody concentrations ≥ 0.1 International unit (IU)/mL | 1 month post third vaccination
  Anti-Tetanus antibodies will be measured by enzyme-linked immunosorbent assay (ELISA).
Number of participants with ≥ 4 fold increase in anti-PT and anti-FHA antibody concentrations (EU/mL) from 1 month pre-dose 1 to 1 month post-dose 3 | I month post dose 3
  Anti-PT and anti-FHA antibodies will be measured by enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Number of participants with anti-Diphtheria antibody concentrations ≥ 0.01 IU/mL and ≥ 0.1 IU/mL International Units (IU)/mL | Day 0 Pre-vaccination
  Anti-Diphtheria antibodies will be measured by a toxin neutralization test
Number of participants with anti-Hepatitis B antibody concentrations ≥ 10 mIU/mL international unit (IU)/mL | Day 0 Pre-vaccination
  Anti-Hepatitis B antibodies will be measured by the commercially available VITROS ECi/ECiQ Immunodiagnostic System using chemiluminescence detection technology
Number of participants with anti Diphtheria antibody concentrations ≥ 0.1 IU/mL International Units (IU)/mL | 1 month post third vaccination
  Anti-Diphtheria antibodies will be measured by a toxin neutralization test
Number of participants reporting solicited injection site and solicited systemic reactions, unsolicited adverse events, and serious adverse events following vaccination with either DTaP-IPV-Hep B-PRP~T combined vaccine or Pentaxim™ and Euvax B® vaccine | Day 0 and up to Day 180 post-vaccination
  Solicited injection site reactions Tenderness, Erythema, and Swelling. Solicited systemic reactions Fever (temperature), Vomiting, Crying abnormal, Drowsiness, Appetite loss, and Irritability.
Number of participants with response to vaccine Pertussis toxoid (PT) and Filamentous Haemagglutinin (FHA) antigens | 1 month post third vaccination
  Vaccine response defined as: Post-dose 3 anti-PT and anti-FHA antibody concentrations in ELISA units (EU)/mL ≥ 4 x Lower Limit of Quantitation (LLOQ) if pre-vaccination concentration is < 4 x LLOQ or ≥ pre-vaccination concentration if pre-vaccination concentrations ≥ 4 x LLOQ

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (9):
- South Korea (9):
  - Daejeon
  - Gyeonggi-do
  - Gyeongsangnam Do
  - Jeollabuk Do
  - Jeonbuk
  - Kangwon Do
  - Kyunggi Do
  - Seoul
  - Suwon Gyeonggi Do

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com